CLINICAL TRIAL: NCT06537375
Title: Use of Intravenous Ketamine in Patients with Severe Chronic Pain Syndromes
Brief Title: Use of Ketamine in Severe Pain Syndromes
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024171
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: Pain, Intractable; Pain, Chronic; Pain Syndrome; Pain Measurement
MeSH Terms: conditions — Pain, Intractable; Chronic Pain; Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ketamine has been shown to have a certain efficiency in chronic pain syndromes. However, it is still not clearly known what is its efficiency and how ketamine is used in real world patients. In this retrospective study, all patients treated with ketamine for chronic pain in our hospital will be reviewed. Patients demographics, pain syndromes as well as outcome criteria will be collected to describe the use of ketamine in pain syndromes.

DETAILED DESCRIPTION:
The American Society of Regional Anesthesia and Pain Medicine, together with the American Academy of Pain and the American Society of Anesthesiologists published a consensus guideline in 2018 on the use of ketamine in chronic pain. A review of medical charts of all patients who received ketamine for chronic pain between january 2010 and june 2024 will be done. Demographic data, detailed pain scores, as well as description of the type of pain will be collected. Ketamine usage will be recorded for the dosage, as well as duration of the treatment. Outcome will be measured by before/after pain scores for neuropathic pain, as well as on a visual analog scale. A more global score (good-medium-no effect) will also be collected to get the patient's impression on their treatment. Concomitant pain medication will be collected.

ELIGIBILITY:
Inclusion Criteria:

- All patients who received ketamine as treatment for a pain syndrome during january 2010 until june 2024 at Erasme University Hospital

Exclusion Criteria:

* Age < 18 years
* Patients who expressed their opposition to the use of their medical data
* incomplete medical chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received ketamine as treatment for a pain syndrome during january 2010 until june 2024 at Erasme University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 6 month
  A scale (good-medium-no effect) of the efficacity of ketamine on their pain syndrome
DN4 | 6 month
  Neuropathic pain scale 4
VAS | 6 month
  Visual analog scale of the pain intensity

SECONDARY OUTCOMES:
Concomitant pain medications | 6 month
  Number of concomitant pain medications used by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital erasme, Brussels, Belgium